CLINICAL TRIAL: NCT01360398
Title: Contribution of Infectious Pathogens to Acute Respiratory Illness in Adults and Elderly
Brief Title: Infectious Pathogens in Acute Respiratory Illness in Adults and Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 114378
Record Dates: First submitted 2011-05-24; First posted 2011-05-25 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Respiratory Disorders
Keywords: pathogen; Chronic Obstructive Pulmonary Disease; Acute Exacerbations of Chronic Obstructive Pulmonary Disease; COPD; respiratory; AECOPD; exacerbation
MeSH Terms: conditions — Respiration Disorders; Pulmonary Disease, Chronic Obstructive | interventions — Blood Specimen Collection; Data Collection

ARMS (1):
- Cohort (Other): COPD male and female patients between 40 and 85 years of age, recruited among the patients of the Southampton General Hospital and referring practices.
  Interventions: Procedure: Blood sample; Procedure: Sputum sample; Procedure: Nasopharyngeal swab; Procedure: Urine sample; Procedure: End tidal breath sample; Other: Data collection; Other: Tests

INTERVENTIONS:
Procedure: Blood sample — Blood samples will be collected from all patients at enrolment, at follow-up visits, at exacerbation visits, and during the final visit.
Procedure: Sputum sample — Sputum will be collected from all patients at enrolment, at monthly follow-up visits, at exacerbation visits, and during the final visit. Sputum will be obtained by spontaneous expectoration or induced by stimulation according to standard methods.
Procedure: Nasopharyngeal swab — Nasopharyngeal swabs will be collected from all patients at enrolment and from a subcohort of 30 patients at monthly follow-up visits and at exacerbation visits during the first year.
Procedure: Urine sample — Urine samples will be taken at enrolment and exacerbation visits from all subjects and from the same subcohort of 30 patients providing nasopharyngeal swabs, at monthly follow-up visits during the first year.
Procedure: End tidal breath sample — Breath samples will be collected from all patients at enrolment, at follow-up visits (monthly), at exacerbation visits, and during the final visit.
Other: Data collection — Patient interview, diary cards review and questionnaires completion
Other: Tests — Urine pregnancy test, chest CT-scan, lung function testing and 6-min walk test

SUMMARY:
The aim of this study is to generate epidemiological data to further explore determinants of Chronic Obstructive Pulmonary Disease (COPD) and the contribution of bacterial and viral pathogens to Acute Exacerbation of COPD (AECOPD) episodes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Male or female subjects between, and including, 40 and 85 years of age, at the time of consent.
* Subjects with confirmed diagnosis of COPD with Forced Expiratory Volume of air expired in 1 second (FEV1) of </=80% of predicted normal and FEV1/Forced expiratory Vital Capacity (FVC)<0.7
* Subjects have moderate, severe, or very severe COPD, according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) staging.
* Subjects have a current or prior history of >/=10 pack-years of cigarette smoking. Former smokers are defined as those who have stopped smoking for at least 6 months. Number of pack years = (number of cigarettes per day/20) x number of years smoked.
* Subjects present a documented history of >/=1 exacerbation requiring antibiotics and/or oral corticosteroids or hospitalization in the previous 12 months.

Exclusion Criteria:

* Subject also has a confirmed diagnosis of asthma, cystic fibrosis, pneumonia risk factors or other respiratory disorders.
* Subjects having undergone lung surgery.
* Subject has a α-1 antitrypsin deficiency as underlying cause of COPD.
* Subject who experienced a moderate or severe COPD exacerbation not resolved at least 1 month prior to enrolment visit and at least 30 days following the last dose of oral corticosteroids.
* Subject using any antibacterial, antiviral or respiratory investigational drug or relevant vaccine up to 30 days prior to the enrolment visit.
* Subject has other conditions that the principal investigator judges may interfere with the study findings. Women who are pregnant or lactating or are planning on becoming pregnant during the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2011-06-30 (Actual); Primary Completion 2014-06-27 (Actual); Study Completion 2014-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bourne S, Cohet C, Kim V, Barton A, Tuck A, Aris E, Mesia-Vela S, Devaster JM, Ballou WR, Clarke SC, Wilkinson T. Acute Exacerbation and Respiratory InfectionS in COPD (AERIS): protocol for a prospective, observational cohort study. BMJ Open. 2014 Mar 7;4(3):e004546. doi: 10.1136/bmjopen-2013-004546. PMID 24607562
- [Background] Mayhew D, Devos N, Lambert C, Brown JR, Clarke SC, Kim VL, Magid-Slav M, Miller BE, Ostridge KK, Patel R, Sathe G, Simola DF, Staples KJ, Sung R, Tal-Singer R, Tuck AC, Van Horn S, Weynants V, Williams NP, Devaster JM, Wilkinson TMA; AERIS Study Group. Longitudinal profiling of the lung microbiome in the AERIS study demonstrates repeatability of bacterial and eosinophilic COPD exacerbations. Thorax. 2018 May;73(5):422-430. doi: 10.1136/thoraxjnl-2017-210408. Epub 2018 Jan 31. PMID 29386298
- [Derived] Budroni S, Taccone M, Stella M, Aprea S, Schiavetti F, Bardelli M, Lambert C, Rondini S, Weynants V, Contorni M, Wilkinson TMA, Brazzoli M, Rossi Paccani S. Cytokine Biomarkers of Exacerbations in Sputum From Patients With Chronic Obstructive Pulmonary Disease: A Prospective Cohort Study. J Infect Dis. 2024 Nov 15;230(5):e1112-e1120. doi: 10.1093/infdis/jiae232. PMID 38836471
- [Derived] Brettoni C, Muzzi A, Rondini S, Weynants V, Rossi Paccani S. Ex-vivo RNA expression analysis of vaccine candidate genes in COPD sputum samples. Respir Res. 2023 Oct 5;24(1):243. doi: 10.1186/s12931-023-02525-z. PMID 37798723
- [Derived] Wilkinson TMA, Van den Steen P, Cheuvart B, Baudson N, Dodet M, Turriani E, Harrington L, Meyer N, Rondini S, Taddei L, Mukherjee P. Seroprevalence of Bordetella pertussis Infection in Patients With Chronic Obstructive Pulmonary Disease in England: Analysis of the AERIS Cohort. COPD. 2021 Jun;18(3):341-348. doi: 10.1080/15412555.2021.1920904. Epub 2021 May 6. PMID 33955798
- [Derived] Malvisi L, Taddei L, Yarraguntla A, Wilkinson TMA, Arora AK; AERIS Study Group. Sputum sample positivity for Haemophilus influenzae or Moraxella catarrhalis in acute exacerbations of chronic obstructive pulmonary disease: evaluation of association with positivity at earlier stable disease timepoints. Respir Res. 2021 Feb 24;22(1):67. doi: 10.1186/s12931-021-01653-8. PMID 33627095
- [Derived] Germovsek E, Ambery C, Yang S, Beerahee M, Karlsson MO, Plan EL. A Novel Method for Analysing Frequent Observations from Questionnaires in Order to Model Patient-Reported Outcomes: Application to EXACT(R) Daily Diary Data from COPD Patients. AAPS J. 2019 Apr 26;21(4):60. doi: 10.1208/s12248-019-0319-9. PMID 31028495
- [Derived] Wilkinson TMA, Aris E, Bourne SC, Clarke SC, Peeters M, Pascal TG, Taddei L, Tuck AC, Kim VL, Ostridge KK, Staples KJ, Williams NP, Williams AP, Wootton SA, Devaster JM. Drivers of year-to-year variation in exacerbation frequency of COPD: analysis of the AERIS cohort. ERJ Open Res. 2019 Feb 25;5(1):00248-2018. doi: 10.1183/23120541.00248-2018. eCollection 2019 Feb. PMID 30815467
- [Derived] Williams NP, Ostridge K, Devaster JM, Kim V, Coombs NA, Bourne S, Clarke SC, Harden S, Abbas A, Aris E, Lambert C, Tuck A, Williams A, Wootton S, Staples KJ, Wilkinson TMA; AERIS Study Group. Impact of radiologically stratified exacerbations: insights into pneumonia aetiology in COPD. Respir Res. 2018 Jul 28;19(1):143. doi: 10.1186/s12931-018-0842-8. PMID 30055608
- [Derived] Wilkinson TMA, Aris E, Bourne S, Clarke SC, Peeters M, Pascal TG, Schoonbroodt S, Tuck AC, Kim V, Ostridge K, Staples KJ, Williams N, Williams A, Wootton S, Devaster JM; AERIS Study Group. A prospective, observational cohort study of the seasonal dynamics of airway pathogens in the aetiology of exacerbations in COPD. Thorax. 2017 Oct;72(10):919-927. doi: 10.1136/thoraxjnl-2016-209023. Epub 2017 Apr 21. PMID 28432209
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 114378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Group: Chronic Obstructive Pulmonary Disease [COPD] diagnosed male and female patients between 40 and 85 years of age, recruited among the patients of the Southampton General Hospital and referring practices, enrolled to generate additional data for further exploration of COPD determinants and the contribution of infectious pathogens to Acute Exacerbation of COPD (AECOPD).
Period: Overall Study
Arm/Group | Total Group
Started | 127
Completed | 105
Not Completed | 22
Not completed — Withdrawal by Subject | 14
Not completed — Other | 7
Not completed — Migrated/moved from study area | 1

BASELINE CHARACTERISTICS:
Arm/Group | Total Group
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Estimated Number of Acute Exacerbation of COPD (AECOPD)
Description: An Acute Exacerbation in a COPD patient is an event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough, and/or sputum production and beyond normal day to day variations, that is acute in onset and may warrant a change in regular medication in a patient with underlying COPD The Means and Confidence Intervals (CI) were estimated using the Negative Binomial model taking into account time to follow up. Estimated exacerbations were presented as mean number of exacerbations per (/) subject/ year.
Time Frame: During year 1
Population: The analyses of AECOPD were performed on the Full cohort, which included all subjects eligible for inclusion based on medical history and study specific procedures defined in the protocol and who completed at least the Day 0 visit.
Measure: Mean (95% Confidence Interval); unit: AECOPD/subject/year
Arm/Group | Total Group
Number analyzed (Participants) | 127
AECOPD/subject/year | 3.04 [2.63 to 3.50]

2. Primary Outcome: Mean Estimated Number of AECOPD With Sputum Containing Bacterial Pathogens
Description: Bacterial pathogens assessed were: Haemophilus influenzae (Hi), Moraxella catarrhalis (Mcat), Steptococcus pneumoniae (Sp), Staphylococcus Aureus (Sta), Pseudomonas aeruginosa (Psa), any or other. For each bacteria, the means and CIs were estimated from Negative Binomial model taking into account the follow up time.Estimated exacerbations were presented as mean number of exacerbations/ subject/ year.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: AECOPD/subject/year
Arm/Group | Total Group
Number analyzed (Participants) | 127
AECOPD/subject/year
  Any | 1.59 [1.30 to 1.95]
  Hi | 1.10 [0.84 to 1.43]
  Mcat | 0.34 [0.24 to 0.48]
  Sp | 0.39 [0.27 to 0.58]
  Sta | 0.16 [0.07 to 0.36]
  Psa | 0.18 [0.09 to 0.35]
  Other | 0.01 [0.00 to 0.06]

3. Primary Outcome: Overall AECOPD Exacerbation Rate for Any and Specific Bacterial Pathogens in Sputum
Description: Bacterial pathogens assessed, by culture, were: Haemophilus influenzae (Hi), Moraxella catarrhalis (Mcat), Streptococcus pneumoniae (Sp), Staphylococcus aureus (Sta), Pseudomonas aeruginosa (Psa), any bacteria or other bacteria. Overall exacerbation rate is the average number of exacerbations for each subject during their time in the study.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Number; unit: AECOPD/subject
Arm/Group | Total Group
Number analyzed (Participants) | 127
AECOPD/subject
  Any Bacteria | 1.48
  Hi | 1.02
  Mcat | 0.31
  Sp | 0.37
  Sta | 0.14
  Psa | 0.17
  Other Bacteria | 0.01

4. Secondary Outcome: Number of Sputum Samples Positive for Specific Pathogens - Any Bacteria and Hi
Description: Sputum samples were tested by bacterial species (any bacteria, Hi, Mcat, Sp, Sta, Psa and other bacteria), or overall and were obtained from culture at each visit (enrollment, any stable visit, any exacerbation visit, any mild exacerbation visit, any moderate exacerbation visit, any severe exacerbation visit). This endpoint presents results for any bacteria and Hi.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Number; unit: sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 127
sputum samples
  Any Bacteria - enrollment | 57
  Any Bacteria - any stable visit | 466
  Any Bacteria - any exacerbation visit | 188
  Any Bacteria - any mild exacerbation visit | 17
  Any Bacteria - any moderate exacerbation visit | 162
  Any Bacteria - any severe exacerbation visit | 9
  Hi - enrollment | 32
  Hi - any stable visit | 287
  Hi - any exacerbation visit | 129
  Hi - any mild exacerbation visit | 11
  Hi - any moderate exacerbation visit | 111
  Hi - any severe exacerbation visit | 7

5. Secondary Outcome: Number of Sputum Samples Positive for Specific Pathogens - Mcat and Sp
Description: Sputum samples were tested by bacterial species (any bacteria, Hi, Mcat, Sp, Sta, Psa and other bacteria), or overall and were obtained from culture at each visit (enrollment, any stable visit, any exacerbation visit, any mild exacerbation visit, any moderate exacerbation visit, any severe exacerbation visit). This endpoint presents results for Mcat and Sp.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Number; unit: sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 127
sputum samples
  Mcat - enrollment | 8
  Mcat - any stable visit | 50
  Mcat - any exacerbation visit | 40
  Mcat - any mild exacerbation visit | 1
  Mcat - any moderate exacerbation visit | 39
  Mcat - any severe exacerbation visit | 0
  Sp - enrollment | 19
  Sp - any stable visit | 177
  Sp - any exacerbation visit | 47
  Sp - any mild exacerbation visit | 6
  Sp - any moderate exacerbation visit | 37
  Sp - any severe exacerbation visit | 4

6. Secondary Outcome: Number of Sputum Samples Positive for Specific Pathogens - Sta, Psa and Other Bacteria
Description: Sputum samples were tested by bacterial species (any bacteria, Hi, Mcat, Sp, Sta, Psa and other bacteria), or overall and were obtained from culture at each visit (enrollment, any stable visit, any exacerbation visit, any mild exacerbation visit, any moderate exacerbation visit, any severe exacerbation visit). This endpoint presents results for Sta, Psa and other bacteria.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Number; unit: sputum samples
Arm/Group | Total Group
Number analyzed (Participants) | 127
sputum samples
  Sta - enrollment | 6
  Sta - any stable visit | 40
  Sta - any exacerbation visit | 18
  Sta - any mild exacerbation visit | 0
  Sta - any moderate exacerbation visit | 18
  Sta - any severe exacerbation visit | 0
  Psa - enrollment | 6
  Psa - any stable visit | 49
  Psa - any exacerbation visit | 21
  Psa - any mild exacerbation visit | 0
  Psa - any moderate exacerbation visit | 19
  Psa - any severe exacerbation visit | 2
  Other bacteria - enrollment | 2
  Other bacteria - any stable visit | 6
  Other bacteria - any exacerbation visit | 1
  Other bacteria - any moderate exacerbation visit | 0
  Other bacteria - any mild exacerbation visit | 1
  Other bacteria - any severe exacerbation visit | 0

7. Secondary Outcome: Mean Number of Days Between 2 Consecutive AECOPDs
Description: The number of days between 2 consecutive exacerbations, as estimated by the investigator, was calculated only whenever the first exacerbation had an end date.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Total Group
Number analyzed (Participants) | 127
Days | 55.5 (53.0)

8. Secondary Outcome: Change From Baseline EXAcerbations of Chronic Pulmonary Disease Tool (EXACT) Scores at Enrollment and Any AECOPD Visit
Description: The exacerbations of chronic pulmonary disease tool version 1.0 (EXACT) is a validated self-administered instrument that evaluates the effects of pharmacologic treatment on acute exacerbations of COPD. Analyses of exacerbations in relation to morning or evening EXACT-PRO e-diaries were presented as follows: descriptive statistics on the EXACT daily scores tabulated at enrolment, at any stable and at any, mild, moderate or severe exacerbation visit. EXACT-PRO contains 14 questions with scores ranging from 0 to 4, where 0= best outcome while 4= worse outcome.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: COPD EXACT Score
Arm/Group | Total Group
Number analyzed (Participants) | 127
COPD EXACT Score
  Enrollment | 0.0 (0.00)
  Any stable visit | -3.0 (9.34)
  Any onset of exacerbation visit | 2.7 (10.24)
  Any onset of mild exacerbation visit | 0.3 (11.16)
  Any onset of moderate exacerbation visit | 2.9 (10.30)
  Any onset of severe exacerbation visit | 2.3 (5.58)

9. Secondary Outcome: Change From Baseline COPD Assessment Test (CAT) Scores at Enrollment and Any AECOPD Visit
Description: The COPD assessment test (CAT) is a validated self-administered instrument designed to provide a simple and reliable measure of health status in COPD patients. Its properties have been shown to be similar to the St George's respiratory questionnaire (SGRQ). The CAT comprises 8 items and has a scoring range of 0-40, 0= most positive answer and 40= most negative answer. In this study, the subjects were to complete the CAT questionnaire every 3 months.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: COPD CAT Score
Arm/Group | Total Group
Number analyzed (Participants) | 127
COPD CAT Score
  Enrollment | 0.0 (0.00)
  Any stable visit | -0.9 (6.04)
  Any onset of exacerbation visit | 4.1 (7.40)
  Any onset of mild exacerbation visit | 0.3 (5.17)
  Any onset of moderate exacerbation visit | 4.3 (7.43)
  Any onset of severe exacerbation visit | 7.2 (8.14)

10. Secondary Outcome: Change From Baseline COPD Nottingham Extended Activities of Daily Living Scale (NEADL) Scores at Enrollment and Any AECOPD Visit
Description: The NEADL assessed (quarterly in the present study) the ease or difficulty in performing extended activities of daily living. The NEADL scale contains 22 items, each measured on a 4-point Likert scale. There are four dimensions: mobility (6 items); kitchen (5 items); domestic (5 items); leisure (6 items). These are summed producing a total score reflecting general functioning. Each of the 22 individual items had 2 possible scores (0 or 1). Therefore, the range of the NEADL score was 0 to 22. Lower scores indicate greater levels of disability while higher scores indicate greater independence.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: NEADL AECOPD scores
Arm/Group | Total Group
Number analyzed (Participants) | 127
NEADL AECOPD scores
  Enrolment | 0.0 (0.00)
  Any stable visit | 6.2 (13.41)
  Any onset of exacerbation visit | 3.2 (12.78)
  Any onset of mild exacerbation visit | 3.8 (8.95)
  Any onset of moderate exacerbation visit | 3.3 (13.18)
  Any onset of severe exacerbation visit | 0 (11.16)

11. Secondary Outcome: Change From Baseline COPD EQ-5D Index and Visual Analogue Scale (VAS) Scores at Enrollment and Any AECOPD Visit
Description: The EQ-5D is an established measure of generic health outcome that provides a simple descriptive profile and a single index value that can be used in clinical and economic evaluation of healthcare and in population surveys. Its current format is 3-level and 5 dimensional (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The EQ-5D index was derived from the ratings recorded every 3 months for each of the five individual items (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The EQ-5D index was 0 (worst health state) to 100 (best health state). The negative numbers presented represent a decrease from baseline values and a worsening of health.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: EQ-5D AECOPD scores
Arm/Group | Total Group
Number analyzed (Participants) | 127
EQ-5D AECOPD scores
  Enrolment | 0.0 (0.00)
  Any stable visit | -1.4 (19.25)
  Any onset of exacerbation visit | -14.8 (20.88)
  Any onset of mild exacerbation visit | -4.3 (18.78)
  Any onset of moderate exacerbation visit | -15.8 (20.44)
  Any onset of severe exacerbation visit | -16.9 (28.42)

12. Secondary Outcome: Number of Subjects Receiving Various Health Care Types During AECOPD
Description: AECOPD health care type included: general practitioners (other than the study doctor), pneumologists, other specialists, hospital emergency department, home care nurses, pulmonary rehabilitation programs and/or nutrition advices.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 108
Participants
  General practitioner - Negative | 82
  General practitioner - Positive | 26
  Pneumologist - Negative | 104
  Pneumologist - Positive | 4
  Other specialist - Negative | 103
  Other specialist - Positive | 5
  Emergency department at the hospital - Negative | 96
  Emergency department at the hospital - Positive | 12
  Nurse home care - Negative | 108
  Pulmonary rehabilitation program - Negative | 98
  Pulmonary rehabilitation program - Positive | 10
  Nutrition Advice - Negative | 107
  Nutrition Advice - Positive | 1

13. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Possibly Related/Linked to Withdrawal
Description: Serious adverse events (SAEs) include medical occur-rences that result in death, are life threatening, require hospitali-zation or prolongation of hospitalization or result in disabil-ity/incapacity.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 127
Participants | 0

14. Secondary Outcome: AECOPD Rate With Overall and Specific Bacterial Pathogens in Sputum , by Polymerase Chain Reaction (PCR) Assay
Description: Bacterial pathogens assessed, by PCR assay were: Hi, Mcat, Sp, Sta, Psa, Streptococcus pyogenes (Spyo) and any bacteria.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Number; unit: AECOPD/subject
Arm/Group | Total Group
Number analyzed (Participants) | 127
AECOPD/subject
  Any Bacteria | 1.61
  Hi | 1.30
  Mcat | 0.47
  Sp | 0.20
  Sta | 0.09
  Psa | 0.14
  Spyo | 0.00

15. Secondary Outcome: AECOPD Rate With Overall and Specific Viral Pathogens in Sputum
Description: Viral pathogens assessed were: respiratory syncytial virus (RSV), parainfluenza virus (PIV), entero rhinovirus (ENV), human metapneumovirus (HMP), influenza virus (INV), adenovirus (ADV), coronavirus (CRV), human bocavirus (HBoV) and any virus.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Number; unit: AECOPD/subject
Arm/Group | Total Group
Number analyzed (Participants) | 127
AECOPD/subject
  Any virus | 0.99
  RSV | 0.02
  PIV | 0.05
  ENV | 0.63
  HMP | 0.05
  INV | 0.06
  ADV | 0.02
  CRV | 0.17
  HBoV | 0.02

16. Secondary Outcome: Mild-AECOPD Rate With Overall and Specific Viral Pathogens in Sputum
Description: Viral pathogens assessed were: respiratory syncytial virus (RSV), parainfluenza virus (PIV), entero rhinovirus (ENV), human metapneumovirus (HMP), influenza virus (INV), adenovirus (ADV), coronavirus (CRV), human bocavirus (HBoV) and any virus. Mild exacerbations were defined as worsening symptoms of COPD that were self-managed by the patient.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Number; unit: AECOPD/subject
Arm/Group | Total Group
Number analyzed (Participants) | 127
AECOPD/subject
  Any Virus | 0.08
  RSV | 0.00
  PIV | 0.02
  ENV | 0.05
  HMP | 0.00
  INV | 0.00
  ADV | 0.00
  CRV | 0.02
  HBoV | 0.00

17. Secondary Outcome: Moderate-AECOPD Rate With Overall and Specific Viral Pathogens in Sputum
Description: Viral pathogens assessed were: respiratory syncytial virus (RSV), parainfluenza virus (PIV), entero rhinovirus (ENV), human metapneumovirus (HMP), influenza virus (INV), adenovirus (ADV), coronavirus (CRV), human bocavirus (HBoV) and any virus. Moderate exacerbations were defined as worsening symptoms of COPD that required treatment with oral corticosteroids and/or antibiotics.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Number; unit: AECOPD/subject
Arm/Group | Total Group
Number analyzed (Participants) | 127
AECOPD/subject
  Any Virus | 0.85
  RSV | 0.02
  PIV | 0.03
  ENV | 0.54
  HMP | 0.04
  INV | 0.06
  ADV | 0.02
  CRV | 0.14
  HBoV | 0.02

18. Secondary Outcome: Severe-AECOPD Rate With Overall and Specific Viral Pathogens in Sputum
Description: Viral pathogens assessed were: respiratory syncytial virus (RSV), parainfluenza virus (PIV), entero rhinovirus (ENV), human metapneumovirus (HMP), influenza virus (INV), adenovirus (ADV), coronavirus (CRV), human bocavirus (HBoV) and any virus. Severe exacerbations were defined as worsening symptoms of COPD that required treatment with in-patient hospitalisation or home care intervention.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Number; unit: AECOPD/subject
Arm/Group | Total Group
Number analyzed (Participants) | 127
AECOPD/subject
  Any Virus | 0.06
  RSV | 0.00
  PIV | 0.00
  ENV | 0.04
  HMP | 0.01
  INV | 0.01
  ADV | 0.00
  CRV | 0.01
  HBoV | 0.00

19. Secondary Outcome: AECOPD Rate With Overall and Specific Bacterial Pathogens in Sputum by Severity
Description: An Acute Exacerbation in a COPD patient is an event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough, and/or sputum production and beyond normal day to day variations, that is acute in onset and may warrant a change in regular medication in a patient with underlying COPD. AECOPD severity was assessed as: any, mild, moderate and severe. Any = any COPD symptom regardless of severity. Mild = Worsening symptoms of COPD that are self-managed by the patient. Moderate = Worsening symptoms of COPD that require treatment with oral corticosteroids and/or antibiotics. Severe = Worsening symptoms of COPD that require treatment with in-patient hospitalisation or home care intervention.
Time Frame: During Year 1
Population: as for outcome 1
Measure: Number; unit: AECOPD/subject
Arm/Group | Total Group
Number analyzed (Participants) | 127
AECOPD/subject
  Any AECOPD | 1.48
  Mild AECOPD | 0.13
  Moderate AECOPD | 1.28
  Severe AECOPD | 0.07

ADVERSE EVENTS:
Time Frame: SAEs during Year 1 of the study period
Description: Other (Non-Serious) Adverse Events were not collected as blood sampling was the only invasive procedure performed.
Arm/Group | Total Group
All-Cause Mortality (participants affected / at risk) | 0/127
Serious Adverse Events (participants affected / at risk) | 0/127
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.